CLINICAL TRIAL: NCT00573313
Title: Effects of SAMe in Patients With Alcoholic Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Abbott (Industry); Joint Clinical Research Center (Other); University of Colorado, Denver (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200311168; R01AA014562 (NIH); NIAAA_HAL-014562 (Other: UC Davis)
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Liver Disease, Alcoholic
Keywords: Alcoholic Liver Disease (ALD); S-adenosylmethionine; SAMe
MeSH Terms: conditions — Liver Diseases, Alcoholic | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-adenosylmethionine (SAMe) (Experimental): Alcoholic liver disease patients receiving S-adenosylmethionine (SAMe)at 400 mg capsule three times daily for 24 weeks
  Interventions: Drug: S-adenosylmethionine
- Sugar pill (Placebo Comparator): ALD subjects receiving Placebo three times daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-adenosylmethionine — Alcoholic liver disease patients received drug at dose of 400 mg three times daily for 24 weeks.
  Arms: S-adenosylmethionine (SAMe)
Drug: Placebo — Alcoholic liver disease patients received identical size and shape sugar pill placebo three times daily for 24 weeks.
  Arms: Sugar pill

SUMMARY:
Prior studies in animal models have established that the pathogenesis of alcoholic liver disease (ALD) is regulated in part by the effects of chronic alcohol abuse on hepatic methionine metabolism. The hypothesis of the clinical study was that provision of the methionine metabolite S-adenosylmethionine (SAM) would correct abnormal hepatic methionine metabolism thereby effectively treating ALD. The two goals of the clinical research were a)to determine the clinical relationship of aberrant hepatic methionine metabolism to ALD by comparisons of patterns of serum methionine metabolites in groups of ALD patients, alcoholics without liver disease, and normal healthy subjects, and b) to determine the treatment effects of SAM on patterns of serum methionine metabolites and on the histopathology and biochemical features of liver injury in ALD patients.

DETAILED DESCRIPTION:
We assessed a total of 297 potential ALD candidates, from whom 40 were enrolled in the study. In addition, we enrolled 26 gender matched active alcohol drinkers without liver disease (AD) and 28 age and gender matched healthy control subjects (HS). Of the original 40 ALD subjects who provided initial enrollment data, 3 declined to proceed with the trial. Therefore, 37 ALD patients were randomized to receive SAM at a dose of 400 mg or placebo three times daily for 24 weeks. However 11 of these dropped out after initial evaluation, leaving 26 ALD patients, 13 in each arm, who completed the 24 week trial.

ELIGIBILITY:
Inclusion Criteria

* ALD) a history of chronic alcoholism according to established AUDIT and WHO criteria with the presence of clinical and laboratory features of established liver disease. Also, willingness to undergo liver biopsies at start and completion of the study, and to comply with study medication or placebo and required clinic visits and blood sampling.
* a history of chronic alcoholism without evidence of liver disease;
* healthy subjects without history of alcoholism or presence of liver disease.

Exclusion Criteria:

* viral Hepatitis B or C
* hemochromatosis
* Wilson Disease
* sclerosing cholangitis
* primary biliary cirrhosis
* other chronic disease
* renal insufficiency

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Halsted, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Result] Medici V, Peerson JM, Stabler SP, French SW, Gregory JF 3rd, Virata MC, Albanese A, Bowlus CL, Devaraj S, Panacek EA, Rahim N, Richards JR, Rossaro L, Halsted CH. Impaired homocysteine transsulfuration is an indicator of alcoholic liver disease. J Hepatol. 2010 Sep;53(3):551-7. doi: 10.1016/j.jhep.2010.03.029. Epub 2010 May 31. PMID 20561703
- [Result] Medici V, Virata MC, Peerson JM, Stabler SP, French SW, Gregory JF 3rd, Albanese A, Bowlus CL, Devaraj S, Panacek EA, Richards JR, Halsted CH. S-adenosyl-L-methionine treatment for alcoholic liver disease: a double-blinded, randomized, placebo-controlled trial. Alcohol Clin Exp Res. 2011 Nov;35(11):1960-5. doi: 10.1111/j.1530-0277.2011.01547.x. PMID 22044287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between July 1, 2005 and June 30, 2009 through the emergency room and clinics of the University of California Davis Health System.
Pre-assignment Details: Three (3) participants with alcoholic liver disease dropped out before randomization. Participants (128) excluded because did not meet recruitment criteria, (105) because had not telephone or other means of contact, or (24) declined to participate.
Groups:
- Healthy: Subjects were enrolled into this arm for baseline measurement only.
- Lifestyle Counseling: Subjects were enrolled into this arm for baseline measurements only.
Period: Overall Study
Arm/Group | S-adenosylmethionine (SAMe) | Healthy | Sugar Pill | Lifestyle Counseling
Started | 18 (Eighteen participants recruited to start.) | 28 | 19 (Nineteen recruited to start.) | 26
Completed | 13 | 28 | 13 | 26
Not Completed | 5 | 0 | 6 | 0
Not completed — Protocol Violation | 5 | 0 | 6 | 0

BASELINE CHARACTERISTICS:
Population: 294 patients were screened of whom 37 were selected for the SAMe v sugar pill trial. Of those excluded, 128 did not meet inclusion criteria, 105 met inclusion criteria but were excluded because of lack of reliable contact information, and 24 subjects declined to participate, leaving 37 subjects, 18 and 19 in each respective group at baseline.
Groups:
- S-adenosylmethionine (SAMe) Treatment: The treatment group received S-adenosylmethionine (SAM) 400 mg three times daily.
- Healthy: Healthy subjects without alcoholism or liver disease.
- Lifestyle Counseling: Active drinkers non liver disease subjects
- Sugar Pill Placebo: The placebo group received a sugar pill identical in appearance that was taken three times daily.
- Total: Total of all reporting groups
Arm/Group | S-adenosylmethionine (SAMe) Treatment | Healthy | Lifestyle Counseling | Sugar Pill Placebo | Total
Number analyzed (Participants) | 18 | 28 | 26 | 19 | 91
Age, Categorical [Count of Participants; unit: Participants] — Baseline age measure
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 17 | 28 | 25 | 19 | 89
    >=65 years | 1 | 0 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 4 | 6 | 26
  Male | 12 | 18 | 22 | 13 | 65
Region of Enrollment [Number; unit: participants]
  United States | 18 | 28 | 26 | 19 | 91

OUTCOME MEASURES:

1. Primary Outcome: Changes in Serum AST Levels
Description: Biochemical values for liver function tests and histopathology scores were obtained at week 0 and 24 of the treatment trial, and changes in each were recorded. Here are reported changes in aspartate transaminase (AST) as representative of all changes. Since only baseline values were obtained in the Healthy and Lifestyle counseling groups, there are no recorded changes in these two groups.
Time Frame: Week 0 to week 24
Population: Analysis of AST values was based on numbers of participants in each group who completed the study. Analysis is pre-specified to apply only to subjects with alcoholic liver disease.
Measure: Median (Full Range); unit: Units per liter (U/L)
Arm/Group | S-adenosylmethionine (SAMe) | Sugar Pill
Number analyzed (Participants) | 13 | 13
Units per liter (U/L) | -13.5 (51.344) [-35 to 156] | -56 (18.243) [-140 to 5]

2. Secondary Outcome: Changes in Serum SAM
Description: We compared serum levels of SAM at time 0 and week 24 of the study in the alcoholic liver disease groups only, since these parameters were measured in the healthy and lifestyle coaching groups only at baseline.
Time Frame: September 2005- June 2009
Population: Whereas 37 subjects started the protocol, due to protocol violation, there remained 26 subjects, 13 in each group, for final analyses. Here are reported changes in AST values to represent all variables.
Measure: Median (Full Range); unit: nmol/liter
Groups:
- Sugar Pill: ALD subjects receiving placebo sugar pill three times daily for 24 weeks.
Arm/Group | S-adenosylmethionine (SAMe) | Sugar Pill
Number analyzed (Participants) | 13 | 13
nmol/liter | 54 (92.535) [-19 to 393] | 7 (150.5) [-261 to 97]
Statistical Analysis 1: Comparison: S-adenosylmethionine (SAMe) vs Sugar Pill; Power calculation indicated that a sample size of 20 subjects per treatment arm would detect differences between groups of 0.9 within-subject standard deviations or higher at 80% power and 5% level of significance; Test type: Superiority or Other; p = 0.36, ANCOVA — The data provided here are for changes in serum AST levels as representative of all clinical laboratory parameters measured; Analysis of covariance controlled for baseline data, e.g. AST; Ratio of Geometric Means at 24 weeks. = 0.1505, 95% CI 2-sided [-0.1853 to 0.4863], Standard Error of Mean 0.1615 — Obtained median values and ranges and log transformations of SD

ADVERSE EVENTS:
Description: Adverse events were only measured in participants with alcoholic liver disease who were randomized to receive intervention.
Arm/Group | S-adenosylmethionine (SAMe) Treatment | Sugar Pill Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 10/18 | 10/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-adenosylmethionine (SAMe) Treatment (N=18) | Sugar Pill Placebo (N=19)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4) — 4 subjects in the SAM group and 4 subjects in the placebo group reported transient diarrhea during the course of the study.
Headache (Nervous system disorders) | 2 (2) | 0 (0) — 2 subjects in SAM group complained of transient headache.
Abdominal bloating (Gastrointestinal disorders) | 3 (3) | 2 (2) — 3 in the SAM group and 4 in the placebo group complained of transient abdominal bloating.
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) — 2 subjects in the placebo group complained of transient nausea
Night sweats, hair loss, xerostomia (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Relatively small numbers of subjects analyzed with 13 each completers in the treatment and placebo groups. Within each group, violation of protocal by resumption of alcohol intake accounted for dropouts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No